CLINICAL TRIAL: NCT07109024
Title: Pilot Diagnostic Feasibility Trial of Resistance Profiling Using Functional Imaging and Next Generation Sequencing of Refractory GIST
Brief Title: Resistance Profiling Using Functional Imaging and Next Generation Sequencing in Refractory Gastrointestinal Stomal Tumors (GIST)
Acronym: PATHFINDERS
Status: Not yet recruiting | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: University Hospital Münster, Insitute of Pathology (Unknown); University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Johanna Falkenhorst, MD, Universität Duisburg-Essen
Other Study IDs: PATHFINDERS; 70116838 (Other Grant/Funding Number: German Cancer Aid (Deutsche Krebshiilfe))
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: GIST; Resistance; Ripretinib; Progression; Imaging
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Tumor Samples (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Generation of a comprehensive and single-lesion resistance profile — AI-supported image analysis of functional imaging (PET-CT) and previous imaging data and specialized molecular methods (next-generation sequencing) will be combined into a comprehensive resistance profile.

SUMMARY:
Gastrointestinal stromal tumors (GIST) are the most common malignant sarcomas of the gastrointestinal tract. Inhibitors of the mutated driver proteins KIT and PDGFRA can temporarily control disseminated GIST disease but cannot cure it. Recently, the investigators were able to elucidate the two main resistance mechanisms-the coexistence of ATP-binding pocket (AP) and activation loop (AL) mutations, as well as AP/AL combination mutations. Determining these resistance factors requires methods that are not yet established in routine clinical practice. The investigators hypothesize that identifying these factors and creating resistance profiles in the context of the anatomical location of metastatic lesions can open up new, clinically relevant therapeutic options, including local therapies. The aim of this project is to evaluate the practicability of these methods in everyday clinical use. An AI-supported image analysis and specialized molecular methods will be combined into a comprehensive resistance profile and will be provided to the treating physicians to potentially guide treatment decisions.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors are among the most common sarcomas and typically harbor activating mutations of the KIT or PDGFR receptor tyrosine kinases [1-3]. While KIT/PDGFRA-directed therapies have revolutionized treatment, most patients eventually progress [4, 5]. Those progressing on the approved last-line therapy (ripretinib or avapritinib) face a dismal outcome with a poor median overall survival of approximately 6 months. The investigators have recently shown that KIT and PDGFRA remain the dominant oncogenic drivers throughout all treatment lines, including in patients failing 4th or later line ripretinib or avapritinib [6, 7]. Strategies that effectively target KIT (and PDGFRA) remain the most promising treatment strategies regardless of treatment line. Our recent findings further deepened our understanding of kinase inhibitor escape which could greatly help to adapt salvage treatments in the future.

Two types of secondary resistance mutations emerge following selective pressure from kinase inhibitors: Mutations involving either the ATP-binding pocket (AP) or the activation loop (AL) of KIT. The investigators have previously shown that sunitinib and ripretinib exhibit a highly differential sensitivity profile with sunitinib being a potent inhibitor of AP mutations and ripretinib being a highly potent inhibitor of AL mutations [6]. A recent substudy of the INTRIGUE trial (2nd-line sunitinib vs ripretinib in GIST) revealed that liquid biopsies can be highly predictive markers of response by determining heterogeneity of secondary resistance [8]. Patients that display secondary resistance mutations restricted to either the AP or the AL subdomain of KIT show marked clinical benefit to a single drug treatment. However, none of these drugs can control both types of mutations at the same time hence AL-mutations are selected for during sunitinib treatment and AP mutations during ripretinib treatment. Knowledge about the status of heterogeneity could inform about the selection of drugs.

In addition, a novel type of resistance, AP/AL mutations, representing compound mutations that involve both the ABP and the AL on the same allele (in cis) were recently described [7]. Next generation sequencing (NGS) panels fail to detect these mutations in clinical practice, as their identification requires allele-specific, long-read sequencing. AP/AL mutations were observed in half of all patients progressing on ripretinib and preclinical models showed that these mutations confer a highly resistant phenotype that cannot be controlled by any approved drug or any drug currently tested in clinical trials. Notably, the same is true in PDGFRA-mutant GIST with the common D842V primary (AL-) mutation where secondary mutations typically result in AP/AL mutations [6]. Local treatments (radiotherapy, surgery, ablation) currently represent the only approach to counter these hyper-resistant clones.

The investigators conclude that two fundamental mechanisms determine resistance in refractory GIST:

1. Intra-patient heterogeneity of secondary resistance defined by the presence of separate clones harboring ATP-binding pocket (AP) and activation loop (AL) mutations which cannot be inhibited by mono-therapy [8]
2. Compound-mutations involving secondary and tertiary mutations that involve the AP and the AL in cis. [6, 7]

The investigators hypothesize that implementing these recent research insights into a resistance profiler could help to develop adaptive treatment strategies in the future, particularly utilizing local treatment approaches, in patients currently lacking other treatment options. This image-based visualization platform aims to integrate longitudinal image analysis, functional imaging at time of inclusion, treatment-related parameters as well as liquid and tumor biopsies. The combined information will provide a visualization of TKI resistance in a more accessible, anatomically annotated way (as opposed to a pure paper-report of multiple biopsies) which will then be provided to a regular sarcoma expert tumorboard

ELIGIBILITY:
Inclusion Criteria:

* Advanced gastrointestinal stromal tumors history of exposure and progression or intolerance to imatinib, sunitinib, regorafenib and ripretinib
* Clinical indication for PET-CT and tumor biopsy (optional) (sarcoma center tumorboard protocol)
* Age 18 years and older
* FFPE tumor tissue available
* Previous imaging studies available (CT/MRI/PET Abdomen, ideally at baseline, best response and progression)
* ECOG ≤ 2
* Progressing tumor lesion(s) of which one is accessible for biopsy

Exclusion Criteria:

* contraindication for systemic TKI treatment
* contraindication for contrast-enhanced both CT and MRI imaging.
* GIST without KIT or PDGFRA mutations
* pregnant or breastfeeding women
* patient that - to the investigator's discretion - are not able or willing to comply with the provided protocol and visit schemes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastrointestinal stromal tumors history of exposure and progression or intolerance to imatinib, sunitinib, regorafenib and ripretinib
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Number of Patients with a PATHFINDER profile categorization within four weeks | 4 weeks

SECONDARY OUTCOMES:
Technical feasibility: Turnaround-time required to provide the individual profile | 4-8 weeks
  Time in days from patient inclusion to final report of the individual profile
Technical Feasibility: Practicality of sample collection | 4-8 weeks
  Number of samples collected (blood, tumor) per patient
Clinical feasibility: Recruitment and retention rate | 3 years
  Numer of patients recruited within two years and percentage of patients completing follow-up according to the protocol.
Clinical feasibility: Adherence to the diagnostic protocol | 2 years
  Percentage of patients in which all diagnostic tests have been successfully performed.
Economic endpoint: Expenses related to the diagnostic test | 3 years
  Material and personal costs per patient
Patient-centered endpoint: Acceptance of creating the profile and its use for therapeutic decisions outside this study | 2-3 years
  Questions will be answered using a Likert Scale (1-10; 1: not satisfied at all - 10: very satisfied) and will be repeated during clinical visits.
  How satisfied are you with the current diagnostic process and the waiting time? How satisfied are you with your current therapy?
Patient-centered endpoint: Quality of life during the evaluation and follow-up period | 3 years
  Repeated quality of life questionnaires at every clinical visit:
  EORTC-QLQ-C30: Quality of life questionnaire of the European Organization for the Research and Treatment of Cancer containing 30 Questions EQ-5D-5L: An EuroQOL questionnaire comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Clinical utility: Ability of test components to determine heterogeneity of resistance and AP/AL mutations (using ctDNA and long-read sequencing) | 2-3 years
  Concordance of ctDNA analysis (liquid biopsy) results with sequencing of tumor tissue and semi-automated radiologic imaging analysis
Clinical utility: Positive-predictive value of longitudinal imaging for AP/AL mutations | 2 years
  Number of patients with tumor biopsies in which a predicted AP/AL mutation was confirmed by tumor mutational analysis.
Clinical utility: Positive-predictive value of ctDNA to predict response to any subsequent treatment | 3 years
  Progression-free survival analysis by mutational subgroups
Outcome of patients progressing on or intolerant to ripretinib: Progression-free survival of subsequent treatment lines | 3 years
  Progression-free survival of subsequent treatment lines
Outcome of patients progressing on or intolerant to ripretinib: Overall survival (starting from time of consent) | 3 years min.
  Overall survival in months
Outcome of patients progressing on or intolerant to ripretinib: Objective response rate to subsequent treatment lines | 3 years
  Radiologic Response (Choi-Criteria)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Essen, Essen
  - University Hospital Schleswig-Holstein, Dpt. of Hematlogy and Oncology, Lübeck

IPD SHARING:
Plan to Share IPD: Undecided